CLINICAL TRIAL: NCT03740152
Title: Transcranial Near-Infrared Light in Healthy Subjects: a Cerebral Blood Flow Study With Diffuse Correlation Spectroscopy
Acronym: NIR-Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Paolo Cassano, Physician, Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002481
Record Dates: First submitted 2017-08-23; First posted 2018-11-14 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Cognitive Change

STUDY DESIGN:
Masking Description: Participant receives all three types of light: continuous, pulse, and sham. They do not know when they receive each type of light, but they do know that they will receive all three.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial Light Therapy (Experimental): All subjects will be administered 1 week of continuous TLT, 1 week of pulsed TLT, and 1 week of sham TLT.
  Interventions: Device: Transcranial Light Therapy

INTERVENTIONS:
Device: Transcranial Light Therapy — Device: LiteCure® The PhotoBioModulation-1000 (TPBM-1000)

SUMMARY:
Transcranial Light Therapy involves non-invasive and invisible beams of light that increase energy metabolism in the brain. Transcranial light therapy has been found to promote brain metabolism. The purpose of the study is:

To asses the change in cerebral blood flow induced by the Transcranial Continuous and Pulse Near-Infrared Light Therapy in healthy subjects.

To correlate with cognitive performance the change in cerebral blood flow induced by the Transcranial Continuous and Pulse Near-Infrared Light Therapy in healthy subjects.

To correlate with skin pigmentation the change in cerebral blood flow induced by the Transcranial Continuous and Pulse Near-Infrared Light Therapy in healthy subjects.

To assess the safety and tolerability of the Transcranial Continuous and Pulse Near-Infrared Light Therapy in healthy subjects

DETAILED DESCRIPTION:
During study visits a clinician applies transcranial light therapy to both sides of a participant's forehead for about 30 minutes. The study involves, 1 screening visit which may last up to 3 hours, 3 transcranial light therapy treatment visits, and 1 posttreatment visit (5 total visits to the Massachusetts General Hospital).

All eligible participants will have 1 visit with continuous light, 1 visit with pulsed light, and 1 visit with sham light. Cerebral blood flow will be measured before and after each light session using DCS-spectroscopy. During sham transcranial light therapy visits, the transcranial light therapy device will not produce near infrared waves (e.g., light energy that cannot penetrate the skin and cranium). The participant will not know which treatment is received at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age at screening will be between 18 and 70 years old (inclusive).
2. Women of child-bearing potential must use a double-barrier method for birth control (e.g. condoms plus spermicide) if sexually active.
3. Subject Informed Consent obtained in writing in compliance with local regulations prior to enrollment into this study.
4. The subject is willing to participate in this study for at least 5 weeks.

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. The subject is on any psychotropic medication.
3. Psychotherapy is exclusionary unless the subject has had at least 8 weeks of treatment prior to the screening visit.
4. Any current psychiatric disorder (per SCID assessment)
5. Substance or alcohol dependence or abuse in the past 6 months.
6. History of a psychotic disorder or psychotic episode (current psychotic episode per SCID assessment).
7. Bipolar affective disorder (per SCID assessment).
8. Unstable medical or neurological illness, defined as any illness which is not well-controlled with standard-of-care medications (e.g., insulin for diabetes mellitus, HCTZ for hypertension).
9. Suicidal or homicidal ideation as determined by SCID screening.
10. The subject has a significant skin condition (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo) on the subject's scalp that is found to be in proximity to any of the procedure sites.
11. The subject has an implant of any kind in the head (e.g. stent, clipped aneurysm, embolised Arteriovenous Malformation (AVM), implantable shunt - Hakim valve).
12. Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment (in US: Visudyne (verteporfin) - for age related macular degeneration; Aminolevulinic Acid- for actinic keratoses; Photofrin (porfimer sodium) - for esophageal cancer, non-small cell lung cancer; Levulan Kerastick (aminolevulinic acid HCl) - for actinic keratosis; 5-aminolevulinic acid (ALA)- for non-melanoma skin cancer)
13. Recent history of stroke (90 days).
14. Personality traits that rend the subject unsuitable for the study, based on the investigators' clinical judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Cassano, M.D., Principal Investigator — Massachusetts General Hospital Center for Anxiety and Traumatic Stress Disorders
Locations (1):
- Massachusetts General Hospital- Center for Anxiety and Traumatic Stress Disorders, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcranial Light Therapy
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transcranial Light Therapy
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Cerebral Blood Flow (Baseline to Week 5)
Description: Measured using Diffuse Correlation Spectroscopy (DCS) signal.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: mm2/s
Arm/Group | Transcranial Light Therapy
Number analyzed (Participants) | 10
mm2/s | 2.15 (1.76)

2. Secondary Outcome: Change in Accuracy on N-Back Task (Baseline to Week 5)
Description: The N-Back task is a measure of working memory. Participants are presented a sequence of stimuli and they must decide if the current stimulus is the same as the one presented 2 trials ago. Accuracy was measured as a percentage of correct to incorrect trials.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: accuracy percentage
Arm/Group | Transcranial Light Therapy
Number analyzed (Participants) | 10
accuracy percentage | -4.49 (20.84)

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: The safety endpoints will evaluate any reported adverse events within one week from each sessions of TLT.
Time Frame: 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Transcranial Light Therapy
Number analyzed (Participants) | 10
Participants | 3

ADVERSE EVENTS:
Time Frame: Collected over course of entire treatment period and follow-up (5 weeks).
Description: There were no participants that had qualities that would make them at risk for serious adverse events or all-cause mortality in this study with this pre-studied advice.
Groups:
- Transcranial Light Therapy Recipients: All participants
Arm/Group | Transcranial Light Therapy Recipients
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Light Therapy Recipients (N=10)
Weakness/fatigue (Psychiatric disorders) | 1 (1)
Trouble concentrating (Psychiatric disorders) | 1 (1)
Blurred vision (Psychiatric disorders) | 1 (1)
Nausea/vomiting (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT03740152/Prot_SAP_000.pdf